CLINICAL TRIAL: NCT06924853
Title: Single-Blind, Randomized, Controlled, Crossover Study of Autologous Platelet Lysate Versus Saline in Adults With Lumbosacral Radiculopathy
Brief Title: Platelet Lysate vs Saline for Lumbosacral Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RGX2025-01
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Lumbosacral Radiculopathy; Lumbar Radiculopathy
Keywords: lumbosacral radiculopathy; lumbosacral radicular pain; lumbar radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Patients are randomized either to active treatment or control group. Patients in control group can crossover to treatment group after 3-month time point.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Lysate (Experimental): Lumbar transforaminal epidural of autologous platelet lysate
  Interventions: Other: Platelet lysate
- Saline (Placebo Comparator): Lumbar transforaminal epidural of saline
  Interventions: Other: Saline control

INTERVENTIONS:
Other: Platelet lysate — The day prior to or the morning of the procedure patient will have their blood drawn by a phlebotomist into 8 yellow top tubes and 1 purple top tube and processed into 5cc PL of which 4cc will be used for treatment and the remaining 1cc will be frozen and used for QC. A lavender top blood tube will be collected and used for quantitative CBC analysis (Beckman Coulter DxH 500 Series). Patient will lie on table prone with a pillow under their abdomen to flatten their L-spine, sterilely prepped and draped. Provider to put patient in conscious sedation to maintain study blinding. The physician will then use a 25-gauge needle under intermittent x-ray visualization to access the TF space. The physician will inject the TF space with x-ray contrast (0.5mL of OMNIPAQUE) to confirm epidural flow. Once flow is confirmed, the physician will inject 4mL of the PL, and 0.5mL of 0.5% ropivacaine into the epidural space at each level of interest. A 0.22 micron filter will be used.
  Arms: Platelet Lysate
Other: Saline control — The day prior to or the morning of the procedure patient will have their blood drawn by a phlebotomist into 8 yellow top tubes and 1 purple top tube and processed into 5cc PL of which 4cc will be used for treatment and the remaining 1cc will be frozen and used for QC. A lavender top blood tube will be collected and used for quantitative CBC analysis; same as active treatment to maintain blinding. Patient will lie on table prone with a pillow under their abdomen to flatten their L-spine, sterilely prepped and draped. Provider to put patient in conscious sedation to maintain study blinding. The physician will then use a 25-gauge needle under intermittent x-ray visualization to access the TF space. The physician will inject the TF space with x-ray contrast (0.5mL of OMNIPAQUE) to confirm epidural flow. (6) Once flow is confirmed, the physician will inject 4mL of sterile saline (0.9%), and 0.5mL of 0.5% ropivacaine into the epidural space at each level of interest.
  Arms: Saline

SUMMARY:
This is a randomized trial to evaluate and compare platelet lysate epidural injection to saline epidural injection for the treatment of lumbar radiculopathy (sciatica).

DETAILED DESCRIPTION:
This single-center, single-blind, randomized-controlled clinical trial will enroll approximately 20 participants, randomized in a 1:1 ratio to receive either autologous PL (N=10) or saline (N=10) epidural injections for patients with lumbar radiculopathy.

Prior to enrollment, patients will undergo evaluation of medical history, back pain history, lumbar examination, radicular symptoms, medication use and review lumbar spine imaging.

Treatment will consist of lumbar transforaminal epidural at affected level/side. On the morning of the procedure, all patients will undergo a blood draw to maintain blinding of study condition. Patients in the active treatment group will receive an epidural injection of platelet lysate. Patients in the control group will receive an epidural injection of saline.

Patients will be blinded to study condition until the 3-month post-treatment follow-up. After completing the 3-month surveys, the patients will be unblinded. Patients that had been in the saline control group will be given the opportunity to cross-over into the active treatment group and re-start study timeline, completing follow-up surveys at 1, 2, 3- and 6- months.

The primary objective of this study is to compare the changes in patient-reported outcomes between the 2 groups (control versus treatment) for leg pain. Secondary objectives include comparing the change scores of other patient reported outcomes of back pain and function at 3-months, as well as continued evaluation of efficacy and durability up to 6-months in active treatment group. Change scores will be calculated by taking the difference between the 3-month scores and the baseline scores. Patients will complete subject-reported clinical questionnaires at pre-treatment, 1-month, 2-months, 3-months, and 6-months (6-m questionnaires only in the active treatment group).

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18-65 years of age, inclusive, at time of signing informed consent
2. At least moderate pain at screening using Patient Global Impression of Severity (PGIS)
3. Diagnosis of lumbosacral radiculopathy (LSR) radiating to or below the knee in a single dermatomal pattern (L4, L5, or S1) with onset of clinical symptoms less than 2 year prior to screening visit
4. Presence of one of the following: a radicular pattern (L4, L5, or S1) of sensory, reflex or strength changes
5. Presence of persistent unilateral radicular pain. Have significant leg pain, numbness, or tingling that causes the patient to alter or change activities.
6. LSR pain with inadequate response to conservative care (non-operative); participants must have tried at least one anti-inflammatory or analgesic medication (for at least 2 weeks at adequate doses) and at least one of the following: Physical therapy, bed rest, chiropractic manipulations, home directed lumbar and/or exercise programs.
7. Lumbar spine MRI images are available after the onset of clinical symptoms and correlate with localization of clinical symptoms. CT is acceptable for patients with contraindication for MRI.
8. Is independent, ambulatory, and can comply with post-treatment evaluations and visits.
9. Voluntary signature of the IRB approved Informed Consent

Exclusion Criteria:

1. Untreated underlying psychological conditions (e.g. depression, chronic pain syndrome, etc.) as a contributor of pain
2. Bleeding disorders
3. Currently taking anticoagulant or immunosuppressive medication
4. Evidence on MRI or CT of recent vertebral fracture or segmental instability (spondylolisthesis)
5. Inflammatory or auto-immune based pathology (e.g. rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout, pseudogout, etc.)
6. Co-existing hip or knee pain localized to the joint structures that may interfere with the participant's ability to participate in the study or interfere with pain assessments
7. Any central canal stenosis with neurogenic claudication (not including foraminal stenosis) with pain present mostly during walking and signs of lumbar stenosis on lumbar spine MRI/CT
8. Has undergone a surgical procedure for back pain (e.g. discectomy, artificial disc replacement, fusion, etc)
9. Presence of spinal cord stimulator
10. Received epidural steroid injection or nerve blocks within the last 2 months
11. Use of chronic opioids
12. Documented history of drug abuse within the last 6 months
13. Use of immunosuppressants, oral or intravenous steroids in the last 3 months
14. Is pregnant
15. Allergy or intolerance to study medication (e.g. lidocaine, etc.)
16. Condition represents a worker's comp case and/or is involved in health-related litigation
17. Presence of clinically significant disease that may interfere with the evaluation of safety and other clinical outcomes in the study
18. Any other condition, that in the opinion of the investigator, would preclude the patient from enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Scale (NPS)-Leg | 3-months
  Difference in Numeric Pain Scale group differences (scale 0-10, where 0=no pain and 10=worst possible pain in regard to leg pain

SECONDARY OUTCOMES:
Numeric Pain Scale (NPS)-Leg | Baseline, 1-month, 2-month, 3-month, 6-month
  Changes in NPS from pre to post treatment; scale ranges from 0-10 where 0=no pain and 10=worst possible pain
Numeric Pain Scale (NPS)-Back | Baseline, 1-month, 2-month, 3-month, 6-month
  Changes in NPS from pre to post treatment; scale ranges from 0-10 where 0=no pain and 10=worst possible pain
Mean modified SANE scores | Baseline, 1-month, 2-month, 3-month, 6-month
  Average SANE scores post-treatment; scores range from 0-100 where 0=no improvement and 100=100% improved
Functional Rating Index (FRI) | Baseline, 1-month, 2-month, 3-month, 6-month
  Changes in FRI from pre to post treatment and between group differences at 3 months; scales 0-100% where 0%=no disability and 100%=very severe disability
Oswestry Disability Index (ODI) | Baseline, 1-month, 2-month, 3-month, 6-month
  Changes in ODI from pre to post and between group differences at 3 months; scales 0-100% where 0%=no disability and 100%=very disabled.
Patient Global Impression of Change (PGIC) | 1-month, 2-month, 3-month, 6-month
  Evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status (From "Very Much Improved" to "Very Much Worse")
Patient Global Impression of Severity (PGIS) | Baseline
  Evaluate the severity of your overall health status (From "None" to "Very Severe"
Incidence rate of adverse events | 1-month, 2-month, 3-month, 6-month
  Incidence of adverse events after treatment
Incidence rate of surgical/other treatment interventions | 1-month, 2-month, 3-month, 6-month
  Incidence of surgical/other treatment interventions after treatment
Pain medications | Baseline and 3-months
  Changes in medications from pre to post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Centeno-Schultz Clinic, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams C, Jerome M, Fausel C, Dodson E, Stemper I, Centeno C. Regenerative Injection Treatments Utilizing Platelet Products and Prolotherapy for Cervical Spine Pain: A Functional Spinal Unit Approach. Cureus. 2021 Oct 8;13(10):e18608. doi: 10.7759/cureus.18608. eCollection 2021 Oct. PMID 34659923
- [Background] Tarulli AW, Raynor EM. Lumbosacral radiculopathy. Neurol Clin. 2007 May;25(2):387-405. doi: 10.1016/j.ncl.2007.01.008. PMID 17445735
- [Background] Tuakli-Wosornu YA, Terry A, Boachie-Adjei K, Harrison JR, Gribbin CK, LaSalle EE, Nguyen JT, Solomon JL, Lutz GE. Lumbar Intradiskal Platelet-Rich Plasma (PRP) Injections: A Prospective, Double-Blind, Randomized Controlled Study. PM R. 2016 Jan;8(1):1-10; quiz 10. doi: 10.1016/j.pmrj.2015.08.010. Epub 2015 Aug 24. PMID 26314234
- [Background] Capelli C, Domenghini M, Borleri G, Bellavita P, Poma R, Carobbio A, Mico C, Rambaldi A, Golay J, Introna M. Human platelet lysate allows expansion and clinical grade production of mesenchymal stromal cells from small samples of bone marrow aspirates or marrow filter washouts. Bone Marrow Transplant. 2007 Oct;40(8):785-91. doi: 10.1038/sj.bmt.1705798. Epub 2007 Aug 6. PMID 17680021
- [Background] Centeno C, Markle J, Dodson E, Stemper I, Hyzy M, Williams C, Freeman M. The use of lumbar epidural injection of platelet lysate for treatment of radicular pain. J Exp Orthop. 2017 Nov 25;4(1):38. doi: 10.1186/s40634-017-0113-5. PMID 29177632